CLINICAL TRIAL: NCT02469012
Title: Evaluation of Quality of Life, Neurocognitive Performance, Fatigue, and Emotional State in HCV Patients Before, During, and in the (Long-term) Follow-up of an IFN-free Antiviral Therapy
Brief Title: Neurocognitive Performance and Emotional State in HCV Patients With IFN-free Antiviral Therapy
Acronym: IFNfreeCOG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Wuerzburg (Other)
Responsible Party: Principal Investigator, Arne Schaefer, PD Dr. Arne Schaefer, University of Wuerzburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 228/14
Record Dates: First submitted 2015-05-05; First posted 2015-06-11 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Hepatitis C, Chronic
Keywords: chronic hepatitis C; antiviral treatment; interferon-free; neurocognitive performance; emotional state; quality of life
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Sofosbuvir; Ribavirin; daclatasvir; ledipasvir, sofosbuvir drug combination; 5-fluorouracil, salicylic acid drug combination; ledipasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IFN-free antiviral treatment (Experimental): Combination #1 or Combination #2 or Combination #3 or Combination #4 or Combination #5
  Interventions: Drug: Combination #1; Drug: Combination #2; Drug: Combination #3; Drug: Combination #4; Drug: Combination #5

INTERVENTIONS:
Drug: Combination #1 — Sofosbuvir + Ribavirin
  Other Names: Sofosbuvir + Ribavirin
Drug: Combination #2 — Sofosbuvir + Daclatasvir
  Other Names: Sofosbuvir + Daclatasvir
Drug: Combination #3 — Sofosbuvir + Daclatasvir + Ribavirin
  Other Names: Sofosbuvir + Daclatasvir + Ribavirin
Drug: Combination #4 — Sofosbuvir + Ledipasvir
  Other Names: Sofosbuvir + Ledipasvir
Drug: Combination #5 — Sofosbuvir + Ledipasvir + Ribavirin
  Other Names: Sofosbuvir + Ledipasvir + Ribavirin

SUMMARY:
The present study evaluates neurocognitive performance as well as measures of mood, quality of life, and fatigue in patients with chronic hepatitis C infection. In a prospective longitudinal study design, included patients are monitored before, during, and in the long-term follow-up of interferon-free antiviral treatment (Sofosbuvir +/-Daclatasvir +/- Ribavirin or Sofosbuvir/Ledipasvir +/- Ribavirin). Main study goals are to compare post therapy results of sustained virologic responders to corresponding pretreatment values as well as to historic interferon-treatment patients without virological response. It is expected that HCV-associated neuropsychiatric symptoms and neurocognitive impairment is - at least in part - reversible by the successful application of modern IFN-free antiviral medication.

DETAILED DESCRIPTION:
Chronic hepatitis C is one of the most frequent infectious diseases worldwide and a major cause of chronic liver disease. At diagnosis, approximately 20 % of patients with chronic hepatitis C already have liver cirrhosis.

Therapy for hepatitis C has meanwhile reached a high level of efficacy and effectiveness: at present, about 90 % of patients treated with a combination of peginterferon alfa, ribavirin and sofosbuvir for up to 12 weeks will reach a sustained loss of hepatitis C virus.

Psychiatric side effects of interferon alfa are well known and may require dose reduction or even premature discontinuation of therapy.

As patients on interferon treatment sometimes report concentration or memory impairment that in some cases interferes considerably with their capacity to manage the requirements of everyday life, the investigators planned and intend to conduct a prospective and longitudinal study evaluating - among other parameters - neurocognitive performance before, during, and after therapy with an antiviral IFN-free therapy.

In previously performed scientific work, the investigators were able to show that interferon-based combination therapy of chronic hepatitis C may cause reversible impairment of neurocognitive performance during treatment period. Moreover, the investigators have recently demonstrated that successful IFN-based antiviral treatment (criterion: SVR, sustained virological response) leads to significant improvement of relevant aspects of attentional and neurocognitive performance. These results indicate that HCV-related neurocognitive impairment is potentially reversible.

Nevertheless, there are still open questions and important issues to be addressed in connection with this field of research, especially regarding several aspects IFN-free antiviral therapy:

Questions to be answered:

* At least 12 months after the end of successfully performed IFN-free antiviral treatment - are psychometrically assessed parameters related to patients' quality of life, fatigue, neurocognitive performance, and mood significantly improved as compared to pretreatment (i.e., baseline) values?
* At least12 months after the end of antiviral treatment, is there a significant difference between patients with and without sustained virological response (special to historical group of IFN-treated patients without a sustained virological response) with respect to neurocognitive performance, emotional state, fatigue and quality of life?
* In the absence of a clinically significant liver damage in patients with chronic hepatitis C - does the mere presence of the hepatitis C virus have any significant influence on neurocognitive or attentional performance? Is it possible to confirm the respective findings yielded in the context of former interferon-based treatment regimens?
* With the current and upcoming IFN-free treatment options - are there still any significant therapy-related changes in symptom areas such as neurocognitive performance, mood or fatigue?

Study Design:

Prospective monocentric study with a longitudinal repeated measures design including hepatitis C patients with indication for standard IFN-free antiviral therapy (sofosbuvir/daclatasvir +/- ribavirin; sofosbuvir/ledipasvir +/- ribavirin) and a long-term follow-up of quality of life, neurocognitive performance, fatigue, and emotional state. Planned sample size: n = 30 hepatitis C patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis C and indication for interferon-free antiviral therapy.
* Written informed consent to study participation, especially to long-term follow-up monitoring of quality of life, emotional state, fatigue, and neurocognitive performance after antiviral treatment.
* Age of study participants: between 18 and 75 years.
* At study entry, all participating patients need to have documented antibodies to HCV and circulating HCV-RNA as measured by reverse-transcription polymerase chain reaction (Cobas Amplicor HCV MonitorTM test, Roche Diagnostics)

Exclusion Criteria:

* Insufficient knowledge of the German language or cognitive impairment (due* to the indispensable application of questionnaires and the TAP, test battery of attentional performance).
* Age under 18 years or over 75 years
* Coinfections such as hepatitis B virus or human immunodeficiency virus
* Severe internal diseases (e.g., cancer, ischemic heart disease, autoimmune disease)
* Major depressive disorder (according to DSM-IV criteria), psychosis, active intravenous drug use or alcohol abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Change in Neurocognitive Performance (computerized TAP - Test Battery for Attentional Performance) | evaluation time points are at baseline, after 4 weeks and 12 weeks of antiviral IFN-free treatment, four weeks and 12 months after the end of antiviral IFN-free therapy
  assessment of changes over treatment time (repeated measures design)

SECONDARY OUTCOMES:
Change in Fatigue (Fatigue Impact Scale - FIS-D, questionnaire) | evaluation time points are at baseline, after 4 weeks and 12 weeks of antiviral IFN-free treatment, four weeks and 12 months after the end of antiviral IFN-free therapy
  assessment of changes over treatment time (repeated measures design)
Change in Health-Related Quality of Life (SF-36, questionnaire) | evaluation time points are at baseline, after 4 weeks and 12 weeks of antiviral IFN-free treatment, four weeks and 12 months after the end of antiviral IFN-free therapy
  assessment of changes over treatment time (repeated measures design)
Change in Emotional State (Hospital Anxiety and Depression Scale HADS, questionnaire) | evaluation time points are at baseline, after 4 weeks and 12 weeks of antiviral IFN-free treatment, four weeks and 12 months after the end of antiviral IFN-free therapy
  assessment of changes over treatment time (repeated measures design)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Kraus, MD, PhD, Principal Investigator — Kreiskliniken Altötting-Burghausen, Burghausen, Germany
Locations (1):
- Kreiskliniken Altötting-Burghausen, Medizinische Klinik II, Burghausen, Bavaria, Germany

REFERENCES:
- [Result] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Result] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Result] Jacobson IM, Gordon SC, Kowdley KV, Yoshida EM, Rodriguez-Torres M, Sulkowski MS, Shiffman ML, Lawitz E, Everson G, Bennett M, Schiff E, Al-Assi MT, Subramanian GM, An D, Lin M, McNally J, Brainard D, Symonds WT, McHutchison JG, Patel K, Feld J, Pianko S, Nelson DR; POSITRON Study; FUSION Study. Sofosbuvir for hepatitis C genotype 2 or 3 in patients without treatment options. N Engl J Med. 2013 May 16;368(20):1867-77. doi: 10.1056/NEJMoa1214854. Epub 2013 Apr 23. PMID 23607593
- [Result] Kraus MR, Schafer A, Wissmann S, Reimer P, Scheurlen M. Neurocognitive changes in patients with hepatitis C receiving interferon alfa-2b and ribavirin. Clin Pharmacol Ther. 2005 Jan;77(1):90-100. doi: 10.1016/j.clpt.2004.09.007. PMID 15637534
- [Result] Kraus MR, Schafer A, Teuber G, Porst H, Sprinzl K, Wollschlager S, Keicher C, Scheurlen M. Improvement of neurocognitive function in responders to an antiviral therapy for chronic hepatitis C. Hepatology. 2013 Aug;58(2):497-504. doi: 10.1002/hep.26229. Epub 2013 Jun 24. PMID 23300053
- [Result] Lawitz E, Mangia A, Wyles D, Rodriguez-Torres M, Hassanein T, Gordon SC, Schultz M, Davis MN, Kayali Z, Reddy KR, Jacobson IM, Kowdley KV, Nyberg L, Subramanian GM, Hyland RH, Arterburn S, Jiang D, McNally J, Brainard D, Symonds WT, McHutchison JG, Sheikh AM, Younossi Z, Gane EJ. Sofosbuvir for previously untreated chronic hepatitis C infection. N Engl J Med. 2013 May 16;368(20):1878-87. doi: 10.1056/NEJMoa1214853. Epub 2013 Apr 23. PMID 23607594
- [Result] Schafer A, Scheurlen M, Kraus MR. [Managing psychiatric side effects of antiviral therapy in chronic hepatitis C]. Z Gastroenterol. 2012 Oct;50(10):1108-13. doi: 10.1055/s-0031-1281682. Epub 2012 Oct 11. German. PMID 23059806
- [Result] Sulkowski MS, Gardiner DF, Rodriguez-Torres M, Reddy KR, Hassanein T, Jacobson I, Lawitz E, Lok AS, Hinestrosa F, Thuluvath PJ, Schwartz H, Nelson DR, Everson GT, Eley T, Wind-Rotolo M, Huang SP, Gao M, Hernandez D, McPhee F, Sherman D, Hindes R, Symonds W, Pasquinelli C, Grasela DM; AI444040 Study Group. Daclatasvir plus sofosbuvir for previously treated or untreated chronic HCV infection. N Engl J Med. 2014 Jan 16;370(3):211-21. doi: 10.1056/NEJMoa1306218. PMID 24428467
- [Result] Alter MJ. The epidemiology of acute and chronic hepatitis C. Clin Liver Dis. 1997 Nov;1(3):559-68, vi-vii. doi: 10.1016/s1089-3261(05)70321-4. PMID 15560058
- [Result] McQuillan GM, Alter MJ, Moyer LA, Lambert SB, Margolis HS. A population-based serologic study of hepatitis C virus infection in the United States. In: Rizetto M, Purcell RH, Gerin JL, Verne G (Eds.) Viral Hepatitis and Liver Disease. Turin, Italy: Edizioni Minerva Medica, 1997
- [Result] Kraus MR, Schafer A, Faller H, Csef H, Scheurlen M. Psychiatric symptoms in patients with chronic hepatitis C receiving interferon alfa-2b therapy. J Clin Psychiatry. 2003 Jun;64(6):708-14. doi: 10.4088/jcp.v64n0614. PMID 12823087
- [Result] Bonaccorso S, Marino V, Biondi M, Grimaldi F, Ippoliti F, Maes M. Depression induced by treatment with interferon-alpha in patients affected by hepatitis C virus. J Affect Disord. 2002 Dec;72(3):237-41. doi: 10.1016/s0165-0327(02)00264-1. PMID 12450640
- [Result] Booth JC, O'Grady J, Neuberger J; Thr Royal College of Physicians of London and the British Society of Gastroenterology. Clinical guidelines on the management of hepatitis C. Gut. 2001 Jul;49 Suppl 1(Suppl 1):I1-21. doi: 10.1136/gut.49.suppl_1.i1. No abstract available. PMID 11413125
- [Result] Dieperink E, Ho SB, Thuras P, Willenbring ML. A prospective study of neuropsychiatric symptoms associated with interferon-alpha-2b and ribavirin therapy for patients with chronic hepatitis C. Psychosomatics. 2003 Mar-Apr;44(2):104-12. doi: 10.1176/appi.psy.44.2.104. PMID 12618532